CLINICAL TRIAL: NCT00005705
Title: Adherence in the Childhood Asthma Management Program
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Other Study IDs: 4489; U01HL048999 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-09

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To evaluate three adherence promoting interventions within the Childhood Asthma Management Program (CAMP), an eight center clinical trial that compared pediatric asthma therapies in children five to twelve years old.

DETAILED DESCRIPTION:
BACKGROUND:

The success of any therapeutic intervention, whether preventive or curative, is ultimately dependent on the individual's adherence to treatment. Unfortunately, the failure of a large percentage of patients to adhere to prescribed medical regimens is a widely recognized and well documented phenomenon. It has been estimated that as many as 50 percent of patients do not take their prescribed medications, and of those remaining, less than two-thirds take their medication as prescribed.

The study was part of a two grant initiative, "Evaluation of Adherence Interventions in Clinical Trials", developed by the Behavioral Medicine Branch staff and the Clinical Trials Branch staff and by members of the Clinical Applications and Prevention Advisory Committee Behavioral Medicine and Prevention Working Groups. The initiative, jointly sponsored by the NHLBI and the National Center for Nursing Research (NCNR), was released in September 1991 and awarded in September 1992.

DESIGN NARRATIVE:

All participants medication adherence was measured by self-report, canister weighing, and with the Nebulizer Chronolog, a microprocessor-based monitor of inhaler adherence that recorded the date and time of each inhaler use. The subjects were assigned to one of three adherence treatment groups; a control condition, an informed condition, and a feedback condition. Adherence outcomes were analyzed with respect to treatment assignment, as well as CAMP measures of asthma morbidity, pulmonary function, medication side effects, psychosocial development, and quality of life. Cost-effectiveness analyses were also conducted.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1996-06 (Actual)

REFERENCES:
- [Background] Wamboldt FS, Bender BG, O'Connor SL, Gavin LA, Wamboldt MZ, Milgrom H, Szefler SJ, Ikle D, Rand C. Reliability of the model MC-311 MDI chronolog. J Allergy Clin Immunol. 1999 Jul;104(1):53-7. doi: 10.1016/s0091-6749(99)70113-2. PMID 10400839